CLINICAL TRIAL: NCT06695975
Title: Occupational Self Analysis in People with a Serious Mental Illness on Occupational Balance, Participation in Meaningful Activities and Life Satisfaction
Brief Title: Occupational Self Analysis in People with a Serious Mental Illness.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Collaborators: Universidad de Burgos (Other); Andaluz Health Service (Other Government)
Responsible Party: Principal Investigator, María Rodríguez Bailón, PHD, University of Malaga
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1792-N-21
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Intervention; Control Condition
Keywords: Occupational self-analysis; Occupational Balance; Occupational Satisfaction; Serious Mental Disorder; meaningful activities

STUDY DESIGN:
Intervention Model Description: The intervention group will participate in te 'Occupational self-analysis' program while the control group will have free time.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Occupational self-analysis (Experimental): "Occupational Self-Analysis" program had the focus on increasing "occupational awareness", making it easier for the participants to analyze their occupations, reflect on whether the activities in which they were involved were meaningful to them and learn about their supports and barriers for occupational participation which allowed modifications to their occupational routines
  Interventions: Behavioral: Occupational self-analysis
- Control group (No Intervention): The control group did not receive any specific intervention, and free time was simply included in their agenda within the Mental Helath Therapeutic Community.

INTERVENTIONS:
Behavioral: Occupational self-analysis — Occupational self analysis program is delivered in group sessions, each session lasting 45 minutes, twice a week. Also Individual sessions are held throughout the program with each participant, with the intention of clarifying certain concepts and resolving specific difficulties that were occurring.The thematic modules worked are 5; occupation-health and difficulty, occupational balance, adaptation strategies to difficulties, social relationships and knowing other realities.
  The methodological strategies used to structure the program were the Model of Human Occupation (MOHO) and the See-Judge-Act methodology
  Arms: Occupational self-analysis

SUMMARY:
In this study we test the efectiveness of an intervention called 'Occupational sefl-analysys' where particiapants are taught to analyze what activities they do and why do they choose those activities. Also they are encouage to reflect about those occupations that don't do but will like to. In case they want to , they can make changes in their occupational routines. After he program we assessed the improvements in life satisfaction, participation in meaningful activities, perception of balance and occupational satisfaction,

DETAILED DESCRIPTION:
The appearance of a mental disorder forces the person to modify their occupational choices and participation, due, among other aspects, to the continuous presence of symptoms and relapses. 'Occupational self-analysis' programs are based on increasing occupational awareness to promote changes in meaningful occupational participation. The objective of this study was to test the effectiveness of the 'Occupational self-analysis' program in people with Serious Mental Disorder specially on life satisfaction, participation in meaningful activities, perception of balance and occupational satisfaction, compared to the standard intervention received in a Therapeutic Community of Mental Health.

The program was implemented for 4 months, twice a week, while the control group received the standard treatment.

Ten people participated in the 'Occupational self-analysis' program. Results show that participants improved their perception of occupational balance and occupational satisfaction, as well as increasing their participation in meaningful activities.

ELIGIBILITY:
Inclusion Criteria:

* Having a serious mental illness
* Living in the Therapeutic Community or attend the device's day program.

Exclusion Criteria:

* Havin Acute psychopathology
* Diagnosis of cognitive impairment
* Dependence or abuse of toxic substances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-28 (Actual)

PRIMARY OUTCOMES:
Satisfaction with Life Scale | From enrollment to the end of treatment at 16 weeks
  It is a self-administered questionnaire that consists of 5 items. It measures the subjective criterion of life satisfaction, with multiple response alternatives ranging between 5 (strongly agree) and 1 (strongly disagree). The score ranges between 5 and 25. The reliability index calculated for the Cronbach's alpha scale indicates that the scale had acceptable internal consistency
Occupational Balance Questionnaire | From enrollment to the end of treatment at 16 weeks
  It consists of a brief self-report questionnaire with 13 items that measure occupational balance. The person has to rate the degree of agreement with each of the statements presented. A 6-point ordinal scale is used ranging from 0 (strongly disagree) to 5 (strongly agree). Thus, the maximum score that can be obtained is 65 points by adding the points for each item which means the greater the occupational balance. The scale, in its Spanish version, has adequate psychometric properties.
Engagement in Meaningful Activities Scale | From enrollment to the end of treatment at 16 weeks
  Is the adaptation to the Spanish context of the "Engagement in Meaningful Activities Survey" (EMAS) (Goldberg et al., 2002) , it is a self-report, it consists of 12 items, developed specifically for people with SMI. Measures the degree of participation in meaningful activities. Items are answered using a 4-point Likert scale ranging from 1 (never) to 4 (always). The score is obtained by the sum of the responses to the 12 items, which ranges from 12-48.
Satisfaction with Daily Occupation - Occupational Balance (SODEO) | From enrollment to the end of treatment at 16 weeks
  It is an instrument based on an interview that consists of 13 items organized under 4 areas: Productivity, Leisure or free time, Housework and Self-care. Evaluates: The number of activities in which the person participates daily, the score can range between 0 and 13. The occupational satisfaction derived from participating in this activity, the participant rates each item ranging from 1 (extremely dissatisfied) to 7 (extremely dissatisfied). satisfied). The satisfaction score can range between 13 and 91. And the perceived occupational balance within each area in terms of doing very little (-2), little (-1), neither much nor little (0), a lot (1) or too much (2). The score range is between -8 and 8.

CONTACTS AND LOCATIONS:
Locations (1):
- Comunidad Terapeutica de salud mental Valme, Dos Hermanas, Sevilla, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fernandez-Solano AJ, Del Bano-Aledo ME, Rodriguez-Bailon M. From thinking to acting: occupational self-analysis tools for use with people with intellectual disability. A pilot study. J Intellect Disabil Res. 2019 Sep;63(9):1086-1096. doi: 10.1111/jir.12621. Epub 2019 Apr 24. PMID 31017354
- [Background] Fernandez-Solano AJ, Del Bano-Aledo ME, Rodriguez-Bailon M. Results of an occupational self-analysis program in people with acquired brain injury. A pilot study. Brain Inj. 2020;34(2):253-261. doi: 10.1080/02699052.2019.1689576. Epub 2019 Nov 15. PMID 31730407